CLINICAL TRIAL: NCT02559570
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Safety and Efficacy Study of a Range of Linaclotide Doses Administered Orally to Children, Ages 6 to 17 Years, Who Fulfill Modified Rome III Criteria for Child/Adolescent Functional Constipation (FC)
Brief Title: A Safety and Efficacy Study of a Range of Linaclotide Doses Administered Orally to Children Ages 6-17 Years Who Fulfill Modified Rome III Criteria for Child/Adolescent Functional Constipation (FC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIN-MD-62
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Functional Constipation in Children Ages 6-17 Years
Keywords: Functional constipation in children; LINZESS
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants aged 6 to 11 or 12 to 17 years received matching placebo linaclotide (LIN), 30 minutes before evening meal, once daily for 4 weeks. Administered as liquid oral solution for participants 6 to 11 years of age and solid oral capsule or liquid oral solution for participants 12 to 17 years of age.
  Interventions: Drug: Placebo
- LIN Dose A (9 ug or 18 ug) (Experimental): Participants aged 6 to 11 years with weight 18 to <35 kg received LIN 9 ug, oral solution, 30 minutes before evening meal, once daily for 4 weeks. Participants aged 6 to 11 years with weight ≥35 kg received LIN 18 ug, oral solution, 30 minutes before evening meal, once daily for 4 weeks. Participants aged 12 to 17 years received LIN 18 ug, oral solution or solid capsules, 30 minutes before evening meal, once daily for 4 weeks.
  Interventions: Drug: LIN Dose A
- LIN Dose B (18 ug or 36 ug) (Experimental): Participants aged 6 to 11 years with weight 18 to <35 kg received LIN 18 ug, oral solution, 30 minutes before evening meal, once daily for 4 weeks. Participants aged 6 to 11 years with weight ≥35 kg received LIN 36 ug, oral solution, 30 minutes before evening meal, once daily for 4 weeks. Participants aged 12 to 17 years received LIN 36 ug, oral solution or solid capsules, 30 minutes before evening meal, once daily for 4 weeks.
  Interventions: Drug: LIN Dose B
- LIN Dose C (36 ug or 72 ug) (Experimental): Participants aged 6 to 11 years with weight 18 to <35 kg received LIN 36 ug, oral solution, 30 minutes before evening meal, once daily for 4 weeks. Participants aged 6 to 11 years with weight ≥35 kg received LIN 72 ug, oral solution, 30 minutes before evening meal, once daily for 4 weeks. Participants aged 12 to 17 years received LIN 72 ug, oral solution or solid capsules, 30 minutes before evening meal, once daily for 4 weeks.
  Interventions: Drug: LIN Dose C
- LIN 145 µg (Experimental): Participants aged 12 to 17 years received LIN 145 ug, oral solution or solid capsules, 30 minutes before evening meal, once daily for 4 weeks.
  Interventions: Drug: LIN 145 µg

INTERVENTIONS:
Drug: Placebo — Participants received matching placebo LIN liquid solution or solid capsules, orally, 30 minutes before evening meal, once daily for 4 weeks.
  Arms: Placebo
Drug: LIN Dose A — Participants received LIN 9 or 18 ug liquid solution or solid capsules, orally, 30 minutes before evening meal, once daily for 4 weeks.
  Other Names: LINZESS
  Arms: LIN Dose A (9 ug or 18 ug)
Drug: LIN Dose B — Participants received LIN 18 or 36 ug liquid solution or solid capsules, orally, 30 minutes before evening meal, once daily for 4 weeks.
  Other Names: LINZESS
  Arms: LIN Dose B (18 ug or 36 ug)
Drug: LIN Dose C — Participants received LIN 36 or 72 ug liquid solution or solid capsules, orally, 30 minutes before evening meal, once daily for 4 weeks.
  Other Names: LINZESS
  Arms: LIN Dose C (36 ug or 72 ug)
Drug: LIN 145 µg — Participants received LIN 145 µg, liquid solution or solid capsules, 30 minutes before evening meal, once daily for 4 weeks.
  Other Names: LINZESS
  Arms: LIN 145 µg

SUMMARY:
The purpose of this study was to evaluate dose response of the safety and efficacy of linaclotide for the treatment of functional constipation (FC), in children age 6-17 years. This study includes up to a 4-week Screening Period, and a 2 to 3-week Pretreatment Period. Participants age 6-11 years will receive oral liquid formulation and participants 12-17 years will receive solid oral capsule or liquid oral solution.

Children ages 6-11 years meeting the entry criteria will be randomized to 1 of 3 doses of linaclotide or placebo for 4 weeks. Children ages 12-17 years meeting the entry criteria will be randomized to 1 of 4 doses of linaclotide or placebo for 4 weeks.

This 4-week study will assess the effects of linaclotide on bowel movement frequency, as well as other bowel symptoms of FC.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs at least 18 kg (kilograms) (39.7 lbs)
* Participant meets modified Rome III criteria for child/adolescent FC: For at least 2 months before the Screening Visit, the participant has had 2 or fewer defecations (with each defecation occurring in the absence of any laxative, suppository, or enema use during the preceding 24 hours) in the toilet per week. In addition, at least once per week, patient meets 1 or more of the following:
* a) History of retentive posturing or excessive volitional stool retention
* b) History of painful or hard bowel movements (BMs)
* c) Presence of a large faecal mass in the rectum
* d) History of large diameter stools that may obstruct the toilet
* e) At least one episode of fecal incontinence per week
* Participant is willing to discontinue any laxatives used before the Pretreatment Visit in favor of the protocol-permitted rescue medicine
* Participant has an average of fewer than 3 spontaneous BMs (SBMs) per week during the 14 days before the randomization day and up to the randomization. An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the BM or the calendar day before the BM
* Participant or participant/guardian/legally authorized representative (LAR) or caregiver is compliant with electronic diary (eDiary) by completing both the morning and evening assessments for 10 out of the 14 days immediately preceding the Randomization Visit

Exclusion Criteria:

* Participant meets Rome III criteria for Child/Adolescent irritable bowel syndrome (IBS): At least once per week for at least 2 months before the Screening Visit, the participant has experienced abdominal discomfort (an uncomfortable sensation not described as pain) or pain associated with 2 or more of the following at least 25% of the time:
* 1. Improvement with defecation
* 2. Onset associated with a change in frequency of stool
* 3. Onset associated with a change in form (appearance) of stool
* Participant reports having more than 1 loose, mushy stool (eDiary-recorded stool consistency of 6 on the Pediatric Bristol Stool Form Scale [p-BSFS]) or any watery stool (eDiary-recorded stool consistency of 7 on the p-BSFS) with any SBM that occurred in the absence of laxative use on the calendar day of the BM or the calendar day before the BM during the 14 days before the randomization day and up to the randomization
* Select medical history or conditions that may be related to other causes of constipation or may interfere with safety and efficacy analyses
* Participant has required manual or hospital-based disimpassion any time prior to randomization
* Participant is unable to tolerate the placebo during the Screening Period

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taryn Weissman, Study Director — Allergan, LLC
Locations (61):
- United States (59):
  - HealthStar Research, LLC, Hot Springs, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - WCCT Global, LLC, Costa Mesa, California
  - Ark Clinical Research, Long Beach, California
  - ACTCA, Inc, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Orange County Research Institute, Ontario, California
  - Center for Clinical Trials, LLC, Paramount, California
  - UCSD Rady Children's Hospital, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Ventura Clinical Trials, Ventura, California
  - Colorado Springs Health Partners, HCP-Clinical Research, LLC, Colorado Springs, Colorado
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Homestead Research Institute, Homestead, Florida
  - RM Medical Research, Homestead, Florida
  - Advanced Medical Research Center, Miami, Florida
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - Children's Center for Digestive Health Care LLC, Atlanta, Georgia
  - Sleepcare Clinical Research Institute, Stockbridge, Georgia
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Kosair Children's Hospital - Pediatric Clinical Research Unit, Louisville, Kentucky
  - Michael W. Simon, MD, PSC, Nicholasville, Kentucky
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - University of Maryland Children's Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Of Minnesota, Minneapolis, Minnesota
  - GI Associates and Endoscopy Center, Jackson, Mississippi
  - Craig A. Speigel, MD, Bridgeton, Missouri
  - Midwest Children Health Research Institute, Lincoln, Nebraska
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Columbia University Medical Center and Morgan Stanley, New York, New York
  - Asheboro Research Associates, Asheboro, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Capital Pediatrics and Adolescent Center PLLC, Raleigh, North Carolina
  - Ohio Pediatric Research Association, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Pediatric Care Specialists, Johnstown, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Montgomery Medical Inc., Smithfield, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Coastal Pediatric Research, Charleston, South Carolina
  - Coastal Pediatrics Associates, Mt. Pleasant, South Carolina
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital/Baylor College Medicine, Houston, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Southwest Children's Research Associates, P.A., San Antonio, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Foothill Family Clinic South / J. Lewis Research, Inc., Salt Lake City, Utah
  - Pediatric Specialists of Virginia, Fairfax, Virginia
  - Virginia Tech Carilion School of Medicine Pediatric, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital of Western Ontario, London, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pediatric participants aged 6 to 11 years were dosed using a weight-based approach. For participants who weighed <35 kg, the doses administered corresponded to about 0.25 to 0.5, 0.5 to 1, or 1 to 2 µg/kg. For participants who weighed ≥35 kg, the doses were not to exceed 0.5, 1, or 2 µg/kg.
Period: Overall Study
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug) | LIN 145 µg
Started | 41 | 36 | 41 | 39 | 16
Completed (Completed = Participants who completed the Treatment period.) | 39 | 34 | 39 | 36 | 14
Not Completed | 2 | 2 | 2 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1
Not completed — Other Miscellaneous Reasons | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants in the randomized population who took at least 1 dose of double-blind study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug) | LIN 145 µg | Total
Number analyzed (Participants) | 41 | 36 | 41 | 39 | 16 | 173
Age, Continuous [Mean (Full Range); unit: years] | 10.7 [6 to 17] | 10.9 [6 to 16] | 11.0 [6 to 17] | 11.3 [6 to 17] | 14.7 [12 to 17] | 11.3 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 25 | 23 | 8 | 93
  Male | 21 | 19 | 16 | 16 | 8 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 29 | 32 | 29 | 11 | 131
  Black or African American | 10 | 7 | 9 | 8 | 4 | 38
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Multiple | 1 | 0 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 12 | 9 | 4 | 40
  Not Hispanic or Latino | 33 | 29 | 29 | 30 | 12 | 133
Spontaneous Bowel Movement (SBM) Frequency Rate [Mean (Full Range); unit: SBMs/week] — SBM was defined as a bowel movement (BM) that occurred in the absence of laxative, suppository, or enema use on the calendar day of the BM or the calendar day before the BM. Participants recorded the occurrence of BMs twice daily at the morning and evening in an electronic diary (eDiary) 14-day prior to randomization and up to randomization.
  SBMs/week | 1.248 [0.00 to 2.90] | 1.462 [0.00 to 2.90] | 1.307 [0.00 to 2.90] | 1.324 [0.00 to 2.90] | 1.810 [0.00 to 4.83] | 1.376 [0.00 to 4.83]

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline (CFB) in 4-week Daytime Abdominal Pain
Description: The abdominal pain score was measured using 5-point scale. Participants answered the questions, How much did your tummy hurt as: 0=none, 1=a tiny bit, 2=a little, 3=some, and 4=a lot. The 4-week daytime abdominal pain was calculated as the average of nonmissing scores in evening eDiary during the Treatment Period with higher value indicating greater symptom severity. Baseline value was the average of non-missing values collected 14 days before randomization. Change from Baseline was calculated as the daytime abdominal pain score during the 4-week treatment period (i.e. average of non-missing daytime scores during 4-week treatment period) - daytime abdominal pain score at baseline. A negative change from Baseline indicates improvement. LSM and SE were calculated using ANCOVA method.
Time Frame: Baseline (14-day prior to randomization) to Week 4
Population: ITT population, all participants who had at least 1 postbaseline entry on BM characteristic assessments that determined occurrences of SBMs (i.e. BM frequency and rescue medication use). No data is reported for LIN 145 μg as it was an exploratory arm group. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 41 | 36 | 41 | 39
score on a scale | -0.291 (0.102) | -0.333 (0.108) | -0.289 (0.102) | -0.171 (0.103)
Statistical Analysis 1: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Test type: Superiority; p = 0.7789, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.042, 95% CI 2-sided [-0.335 to 0.252], Standard Error of Mean 0.149 — ANCOVA model was applied with treatment arm groups (linaclotide doses A, B, and C, and placebo) and age group (6 to 11 years of age and 12 to 17 years of age) as factors and baseline value as covariate
Statistical Analysis 2: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Test type: Superiority; p = 0.9930, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.001, 95% CI 2-sided [-0.282 to 0.284], Standard Error of Mean 0.143 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Test type: Superiority; p = 0.4107, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.120, 95% CI 2-sided [-0.167 to 0.408], Standard Error of Mean 0.146 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline (CFB) in 4-week Overall Spontaneous Bowel Movement (SBM) Frequency Rate During the Treatment Period
Description: SBM was defined as a BM that occurred in the absence of laxative, suppository, or enema use on the calendar day of the BM or the calendar day before the BM. SBM rate was defined as SBMs/week during the 4-week Treatment period. Participants recorded the occurrence of BMs and use of rescue medication, morning and evening, daily in an eDiary since pretreatment period. The SBM frequency rate (SBMs/week) during the analysis period for each participant were calculated as [(total number of SBMs in the analysis period/number of days in the analysis period)*7]. Baseline value was based on values collected 14 days before randomization up to randomization. Change from Baseline was calculated as the SBM frequency rate during the 4-week treatment period - SBM frequency rate at baseline. A positive change from Baseline indicates improvement. Least squares mean (LSM) and standard error (SE) were calculated using analysis of covariance (ANCOVA) method.
Time Frame: Baseline (14-day prior to randomization and up to randomization) to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: SBMs/week
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 41 | 36 | 41 | 39
SBMs/week | 2.000 (0.394) | 1.412 (0.422) | 1.814 (0.397) | 2.364 (0.403)
Statistical Analysis 1: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Test type: Superiority; p = 0.3097, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.588, 95% CI 2-sided [-1.729 to 0.552], Standard Error of Mean 0.577 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Test type: Superiority; p = 0.7384, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.186, 95% CI 2-sided [-1.286 to 0.913], Standard Error of Mean 0.557 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Test type: Superiority; p = 0.5188, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.364, 95% CI 2-sided [-0.748 to 1.477], Standard Error of Mean 0.563 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline (CFB) in 4-week Stool Consistency
Description: Participants used 7-point pediatric Bristol Stool Form (p-BSFS) scale to rate stool consistency for each BM in morning and evening eDiary where 1=small hard lumps or balls like pebbles,2=fat sausage shape but lumpy and hard,3=a sausage but with cracks on it,4=sausage or snake, smooth and soft,5=chicken nuggets, soft smooth blobs,6=oatmeal, fluffy mushy pieces,7=milkshake, watery. Scores in 4-week treatment period were calculated by 2 approaches-1) following derivation similar in earlier adult studies, mean of participants non-missing, SBM associated p-BSFS scores during 4-week treatment period (adult derivation),2) observed weighted average of daily p-BSFS scores during that period. Daily p-BSFS score was average of non-missing morning and/or evening assessments of p-BSFS score from SBMs reported by participants on that specific day. Baseline value was based on values collected 14 days before randomization up to randomization. LSM and SE were calculated using ANCOVA method.
Time Frame: Baseline (14-day prior to randomization and up to randomization) to Week 4
Population: ITT population-participants who had at least 1 postbaseline entry on BM characteristic that determined occurrences of SBMs (BM frequency and rescue medication use). No data is reported for LIN 145 μg as it was exploratory arm group. Observed-cases approach used. Overall number of participants analyzed = who had data at Baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 34 | 32 | 34 | 34
score on a scale
  CFB at Week 4 (Adult derivation) | 0.690 (0.174) | 0.641 (0.177) | 0.652 (0.174) | 1.046 (0.172)
  CFB at Week 4 (Weighted average) | 0.668 (0.167) | 0.606 (0.170) | 0.594 (0.166) | 0.930 (0.165)
Statistical Analysis 1: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Adult derivation; Test type: Superiority; p = 0.8426, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.050, 95% CI 2-sided [-0.543 to 0.444], Standard Error of Mean 0.249 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Adult derivation; Test type: Superiority; p = 0.8770, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.038, 95% CI 2-sided [-0.525 to 0.448], Standard Error of Mean 0.246 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Adult derivation; Test type: Superiority; p = 0.1502, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.356, 95% CI 2-sided [-0.131 to 0.842], Standard Error of Mean 0.246 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Weighted average; Test type: Superiority; p = 0.7949, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.062, 95% CI 2-sided [-0.535 to 0.410], Standard Error of Mean 0.239 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Weighted average; Test type: Superiority; p = 0.7543, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.074, 95% CI 2-sided [-0.540 to 0.392], Standard Error of Mean 0.235 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Weighted average; Test type: Superiority; p = 0.2676, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.262, 95% CI 2-sided [-0.204 to 0.728], Standard Error of Mean 0.235 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline (CFB) in 4-week of Severity of Straining
Description: Severity of straining was scored on 5-point scale for question-When you pooped, how hard did you push? The score ranges from 0= not hard at all,1= I pushed a tiny bit hard,2= I pushed a little hard,3= I pushed hard,4= I pushed very hard with higher scores indicating more severe straining. Participants recorded degree of straining for each BM in morning and evening eDiary. Data was derived as adult derivation and weighted average. Scores during 4-week treatment period were calculated following two approaches - (1) following derivation similar in earlier adult studies, as mean of participant's non-missing, SBM associated straining scores during 4-week treatment period (adult derivation) and (2) as observed weighted average of daily straining scores during that period. Daily straining score was the average of non-missing morning and/or evening assessments of straining score from the SBMs reported by the participants on that specific day. LSM and SE were calculated using ANCOVA method.
Time Frame: Baseline (14-day prior to randomization and up to randomization) to Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 34 | 32 | 34 | 34
score on a scale
  CFB at Week 4 (Adult derivation) | -0.657 (0.145) | -0.710 (0.150) | -0.778 (0.147) | -0.893 (0.145)
  CFB at Week 4 (Weighted average) | -0.656 (0.143) | -0.710 (0.149) | -0.769 (0.145) | -0.855 (0.143)
Statistical Analysis 1: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Adult derivation; Test type: Superiority; p = 0.7997, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.053, 95% CI 2-sided [-0.465 to 0.359], Standard Error of Mean 0.208 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Adult derivation; Test type: Superiority; p = 0.5602, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.121, 95% CI 2-sided [-0.530 to 0.288], Standard Error of Mean 0.207 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Adult derivation; Test type: Superiority; p = 0.2529, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.236, 95% CI 2-sided [-0.641 to 0.170], Standard Error of Mean 0.205 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Weighted average; Test type: Superiority; p = 0.7923, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.054, 95% CI 2-sided [-0.461 to 0.352], Standard Error of Mean 0.206 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Weighted average; Test type: Superiority; p = 0.5802, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.113, 95% CI 2-sided [-0.517 to 0.290], Standard Error of Mean 0.204 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Weighted average; Test type: Superiority; p = 0.3263, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.199, 95% CI 2-sided [-0.600 to 0.201], Standard Error of Mean 0.202 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline (CFB) in 4-week Abdominal Bloating Daytime Symptoms Based on Evening Assessment
Description: Participants recorded their assessment of abdominal bloating in the evening eDiary. Participants answered the question: How big and full did your tummy feel? on a scale, where: 0=none, 1=a tiny bit, 2=a little, 3=medium or 4=very, with a higher score indicating more severe bloating. Baseline value was the average of values collected 14 days before randomization. The 4-week daytime abdominal bloating symptoms were calculated as the average of non-missing scores reported in the evening eDiary during the treatment period. Change from Baseline was calculated as the 4-week daytime abdominal bloating score during the treatment period - daytime abdominal bloating score at baseline. A negative change from Baseline indicates improvement. LSM and SE were calculated using ANCOVA method.
Time Frame: Baseline (14-day prior to randomization) to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 41 | 36 | 41 | 39
score on a scale | -0.314 (0.104) | -0.266 (0.110) | -0.287 (0.104) | -0.275 (0.105)
Statistical Analysis 1: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Test type: Superiority; p = 0.7507, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.048, 95% CI 2-sided [-0.252 to 0.349], Standard Error of Mean 0.152 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Test type: Superiority; p = 0.8505, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.028, 95% CI 2-sided [-0.262 to 0.317], Standard Error of Mean 0.146 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Test type: Superiority; p = 0.7933, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.039, 95% CI 2-sided [-0.254 to 0.332], Standard Error of Mean 0.149 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline (CFB) in 4-week Overall Complete Spontaneous Bowel Movement Frequency Rate (CSBM/Week) During the Treatment Period
Description: SBM was defined as a BM that occurred in the absence of laxative, suppository, or enema use on the calendar day of the BM or the calendar day before the BM. A CSBM was an SBM that was associated with a sense of complete evacuation. Participants recorded their assessment of the sensation of incomplete evacuation for each BM in the morning and evening eDiary. The 4-week overall CSBM frequency rate was calculated as [total number of CSBMs in the analysis period/number of days in the analysis period]*7). Baseline value was based on values collected 14 days before randomization and up to randomization. Change from Baseline was calculated as the CSBM frequency rate during the 4-week treatment period - CSBM frequency rate at baseline. A positive change from Baseline indicates improvement. LSM and SE were calculated using ANCOVA method.
Time Frame: Baseline (14-day prior to randomization and up to randomization) to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: CSBMs/week
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 41 | 36 | 41 | 39
CSBMs/week | 1.240 (0.308) | 0.815 (0.328) | 1.005 (0.309) | 1.320 (0.314)
Statistical Analysis 1: Comparison: Placebo vs LIN Dose A (9 ug or 18 ug); Test type: Superiority; p = 0.3461, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.425, 95% CI 2-sided [-1.313 to 0.463], Standard Error of Mean 0.450 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs LIN Dose B (18 ug or 36 ug); Test type: Superiority; p = 0.5892, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = -0.235, 95% CI 2-sided [-1.095 to 0.624], Standard Error of Mean 0.435 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs LIN Dose C (36 ug or 72 ug); Test type: Superiority; p = 0.8560, ANCOVA; ANCOVA model estimates/t-tests comparing specified treatment groups, controlling for age group and baseline value; Least Squares Mean Difference = 0.080, 95% CI 2-sided [-0.789 to 0.949], Standard Error of Mean 0.440 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in 4-week Fecal Incontinence Daytime Symptoms Based on Evening Assessment
Description: Participants recorded the presence of incontinence episodes in daytime daily since pre-treatment period (14-day prior to randomization) in the evening eDiary for participants randomized following protocol amendment #3. The 4-week daytime fecal incontinence was calculated as the mean of non-missing participant scores reported in the evening eDiary during the Treatment Period. Baseline value was the average of values collected 14 days before randomization. Change from Baseline was calculated as the 4-week fecal incontinence daytime symptoms during the treatment period - fecal incontinence daytime symptoms at baseline. A negative change from Baseline indicates improvement.
  No data is reported for LIN 145 μg as it was an exploratory arm group.
Time Frame: Baseline (14-day prior to randomization) to Week 4
Population: Participants from ITT population included all participants who had at least 1 postbaseline entry on BM characteristic assessments that determined occurrences of SBMs (i.e. BM frequency and rescue medication use) who were randomized following the implementation of fecal incontinence assessment in the protocol (amendment #3).
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug)
Number analyzed (Participants) | 11 | 9 | 13 | 10
incontinence episodes | -0.028 (0.081) | -0.025 (0.083) | -0.009 (0.067) | 0.170 (0.298)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to Day 30 after the last dose for serious adverse events (SAEs) and from first dose up to Day 1 after the last dose for other adverse events
Description: Safety population included all participants in the randomized population who took at least 1 dose of double-blind study treatment.
Arm/Group | Placebo | LIN Dose A (9 ug or 18 ug) | LIN Dose B (18 ug or 36 ug) | LIN Dose C (36 ug or 72 ug) | LIN 145 µg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/36 | 0/41 | 0/39 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/36 | 0/41 | 0/39 | 1/16
Other Adverse Events (participants affected / at risk) | 3/41 | 1/36 | 3/41 | 10/39 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | LIN Dose A (9 ug or 18 ug) (N=36) | LIN Dose B (18 ug or 36 ug) (N=41) | LIN Dose C (36 ug or 72 ug) (N=39) | LIN 145 µg (N=16)
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | LIN Dose A (9 ug or 18 ug) (N=36) | LIN Dose B (18 ug or 36 ug) (N=41) | LIN Dose C (36 ug or 72 ug) (N=39) | LIN 145 µg (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Viral sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT02559570/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT02559570/SAP_001.pdf